CLINICAL TRIAL: NCT02483637
Title: A Prospective Safety and Feasibility Study of the RejuvenAir™ System Metered Cryospray Therapy for Chronic Bronchitis Patients
Brief Title: Safety and Feasibility Study of Rejuvenair™ for Treating Chronic Bronchitis Patients
Acronym: Feasibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CSA Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 012
Record Dates: First submitted 2015-06-25; First posted 2015-06-29 (Estimated); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Bronchitis, Chronic; Cryotherapy Effect
Keywords: spray cryotherapy; cryotherapy; chronic bronchitis; airflow restrictions
MeSH Terms: conditions — Bronchitis, Chronic

STUDY DESIGN:
Intervention Model Description: RejuvenAir
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RejuvenAir (Experimental): RejuvenAir treatment of the right lower lobe and right main stem bronchus. Each MCS will be tailored to the bronchial area undergoing treatment and the amount of liquid nitrogen delivered will vary depending on the airway diameter.
  Interventions: Device: RejuvenAir

INTERVENTIONS:
Device: RejuvenAir — Device: RejuvenAir

SUMMARY:
This study evaluates the safety of RejuvenAir Cryospray therapy to treat symptomatic chronic bronchitis patients with airflow restrictions.

DETAILED DESCRIPTION:
Prospective, open label, single arm study with sequential accrual of subjects with known chronic bronchitis. There are two phases to this study. Phase A will enroll up to 12 subjects and will treat a single lobe to assess safety, feasibility and histology/immunology. After review of the data by the Data Safety Monitoring Board, Phase B of the study would begin. In Phase B of the study, Phase A subjects would have their remaining two lobes treated. In addition up to 24 subjects will be enrolled and will have all upper and lower lobes treated to assess safety, feasibility and immunology.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥40 to ≤75 years of age.
* Subject is able to read, understand, and sign a written Informed Consent in order to participate in the study.
* Subject agrees to continue maintenance pulmonary/COPD medications for the duration of the study.
* Diagnosis of chronic bronchitis (CB) and chronic obstructive pulmonary disease (COPD) for a minimum of two years. (Chronic Bronchitis is defined clinically as chronic productive cough for 3 months in each of 2 successive years in a patient in whom other causes of productive cough have been excluded.)
* Pre-procedure post bronchodilator FEV1 of greater than or equal to 30% and less than or equal to 80% of predicted within 3 months of enrollment.
* Smoking history of at least 10 pack years.
* Non-smoking for a minimum of 6 months prior to consent and agrees to continue not smoking for the duration of the study.
* Subject is able to adhere to and undergo 3 (4 if in Phase A) bronchoscope procedures that includes lung biopsies and multiple MCS treatments in the opinion of the investigator

Exclusion Criteria:

* Subject has had an acute pulmonary infection or pneumonia within prior 6 weeks of study bronchoscopy.
* Subject has had a CB and/or COPD exacerbation (requiring steroids and/or antibiotics) within 6 weeks prior to study bronchoscopy, as defined by their treating physician
* Subject has clinically significant bronchiectasis or other respiratory disease other than chronic bronchitis and COPD.
* Diagnosis of asthma with an onset before 30 years of age
* Subject has bullous emphysema characterized as large bullae >30 millimeters on CT.
* Subject has had a transplant.
* Subject has the inability to walk >140 meters
* Subject has PaC02 >8kPa, or a PaO2<7kPa at room air.
* Subject has a RVSP >45mmHg or a LVEF<45% on 2D-cardiac echo.
* Subject has undergone lung surgery: pneumonectomy, lobectomy, bullectomy, lung volume reduction surgery
* Subject has had a prior lung device procedure, including emphysema stent(s) implanted, lung coils, valves, lung denervation or other devices for emphysema.
* Subject is unable to temporarily discontinue use of anticoagulant therapy:

warfarin, Coumadin, LMWH, heparin, clopidogrel (or equal)

* Subject is on >10 mg of prednisolone/day.
* Subject has a serious medical condition, such as: uncontrolled congestive heart failure, uncontrolled angina, myocardial infarction in the past year, renal failure, liver disease, cerebrovascular accident within the past 6 months, uncontrolled diabetes, hypertension, autoimmune disease or uncontrolled gastric reflux
* Subject is pregnant, nursing, or planning to get pregnant during study duration.
* Subject has received chemotherapy within the past 6 months or is expected to receive chemotherapy during participation in this study.
* Subject is or has been in another clinical investigational study within 6 weeks of baseline.
* Subject has known sensitivity to medication required to perform bronchoscopy (such as lidocaine, atropine, and benzodiazepines).
* Subject has been in another clinical investigational study within 6 weeks of baseline.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02; Primary Completion 2019-05 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Adverse and Serious Adverse Events | Change from Baseline to 3-Months Following Completion of Treatments
  Number of subjects with treatment emergent adverse events. Observed rates and two-sided 95% exact confidence interval will be calculated for AE rates and SAE rates overall and for organ class.
Ability to Complete all 3 MCS Treatments | Change from Baseline to 3-Months Following Completion of Treatments
  Number of subjects completing all 3 treatments.
Patient Reported Outcome Instrument: St. George's Respiratory Questionnaire (SGRQ) | Change from Baseline to 3-Months Following Completion of Treatments
  Scale is 0-100; a higher score is worse

SECONDARY OUTCOMES:
Spirometry Testing | Change from Baseline to 3-Months, 1 year, 2 year and 3 year Following Completion of Treatments
  FEV1, FEV1/FVC, VC, FIV1
6 Minute Walk Test | Change from Baseline to 3-Months, 1 year, 2 year and 3 year Following Completion of Treatments
  Number of meters walked in six minutes
Leicester Cough Questionnaire (LCQ) | Change from Baseline to 3-Months, 1 year, 2 year and 3 year Following Completion of Treatments
  The total score range is 19-133; a higher score is better.
COPD Assessment Test (CAT) | Change from Baseline to 3-Months, 1 year, 2 year and 3 year Following Completion of Treatments
  The total score range is 0-40; a higher score is worse
Visual Analog Scale (VAS) | Change from Baseline to 3-Months, 1 year, 2 year and 3 year Following Completion of Treatments
  The total score range is 0-100; a higher score is worse
Modified Medical Research Council (mMRC) | Change from Baseline to 3-Months, 1 year, 2 year and 3 year Following Completion of Treatments
  The total score range is 0-4; a higher score is worse

OTHER OUTCOMES:
Exacerbation Rate | Change from Baseline to 3-Months, 1 year, 2 year and 3 year Following Completion of Treatments
  Annualized exacerbation rates
Airway Wall Thickness Using HRCT | Change from Baseline to 3-Months, 1 year, 2 year and 3 year Following Completion of Treatments
  Lumen radius in mm.
Plasma Fibrinogen | Change from Baseline to 3-Months, 1 year, 2 year and 3 year Following Completion of Treatments
  150-400mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Heather Nigro, Study Director — CSA Medical
Locations (3):
- St. Paul's Hospital, Vancouver, British Columbia, Canada
- University Medical Center Groningen, Groningen, Netherlands
- Chelsea and Westminster Hosptial/Royal Brompton Hosptial, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thompson AB, Daughton D, Robbins RA, Ghafouri MA, Oehlerking M, Rennard SI. Intraluminal airway inflammation in chronic bronchitis. Characterization and correlation with clinical parameters. Am Rev Respir Dis. 1989 Dec;140(6):1527-37. doi: 10.1164/ajrccm/140.6.1527. PMID 2604284
- [Background] Innes AL, Woodruff PG, Ferrando RE, Donnelly S, Dolganov GM, Lazarus SC, Fahy JV. Epithelial mucin stores are increased in the large airways of smokers with airflow obstruction. Chest. 2006 Oct;130(4):1102-8. doi: 10.1378/chest.130.4.1102. PMID 17035444
- [Background] Ramos FL, Krahnke JS, Kim V. Clinical issues of mucus accumulation in COPD. Int J Chron Obstruct Pulmon Dis. 2014 Jan 24;9:139-50. doi: 10.2147/COPD.S38938. eCollection 2014. PMID 24493923
- [Background] Godwin BL, Coad JE, "Healing responses following cryothermic and hyperthermic tissue ablation. " SPIE Proceedings 2009: Volume 7181, p1-9
- [Background] Sciurba FC, Ernst A, Herth FJ, Strange C, Criner GJ, Marquette CH, Kovitz KL, Chiacchierini RP, Goldin J, McLennan G; VENT Study Research Group. A randomized study of endobronchial valves for advanced emphysema. N Engl J Med. 2010 Sep 23;363(13):1233-44. doi: 10.1056/NEJMoa0900928. PMID 20860505
- [Background] Shah PL, Zoumot Z, Singh S, Bicknell SR, Ross ET, Quiring J, Hopkinson NS, Kemp SV; RESET trial Study Group. Endobronchial coils for the treatment of severe emphysema with hyperinflation (RESET): a randomised controlled trial. Lancet Respir Med. 2013 May;1(3):233-40. doi: 10.1016/S2213-2600(13)70047-X. Epub 2013 Apr 23. PMID 24429129
- [Background] Gibson PG. Cough is an airway itch? Am J Respir Crit Care Med. 2004 Jan 1;169(1):1-2. doi: 10.1164/rccm.2310009. No abstract available. PMID 14695099
- [Background] Jeffery P, Holgate S, Wenzel S; Endobronchial Biopsy Workshop. Methods for the assessment of endobronchial biopsies in clinical research: application to studies of pathogenesis and the effects of treatment. Am J Respir Crit Care Med. 2003 Sep 15;168(6 Pt 2):S1-17. doi: 10.1164/rccm.200202-150WS. No abstract available. PMID 14555461
- [Background] Pulmonary Physiology, Levitzky M. 7th ed. 2007, The McGraw-Hill Companies
- [Background] Smith BM, Hoffman EA, Rabinowitz D, Bleecker E, Christenson S, Couper D, Donohue KM, Han MK, Hansel NN, Kanner RE, Kleerup E, Rennard S, Barr RG. Comparison of spatially matched airways reveals thinner airway walls in COPD. The Multi-Ethnic Study of Atherosclerosis (MESA) COPD Study and the Subpopulations and Intermediate Outcomes in COPD Study (SPIROMICS). Thorax. 2014 Nov;69(11):987-96. doi: 10.1136/thoraxjnl-2014-205160. Epub 2014 Jun 13. PMID 24928812
- [Derived] Agrawal A. Interventional Pulmonology: Diagnostic and Therapeutic Advances in Bronchoscopy. Am J Ther. 2021 Feb 9;28(2):e204-e216. doi: 10.1097/MJT.0000000000001344. PMID 33590989